CLINICAL TRIAL: NCT03806543
Title: The Influencing Factors of Vancomycin Trough Level and the Rate Achieving the Target Trough Level in Critically Ill Patients: A Retrospective Observational Study
Brief Title: The Influencing Factors of Vancomycin Trough Level and the Rate Achieving the Target Trough Level
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Other Study IDs: 2018ZDSYLL117-P01
Record Dates: First submitted 2018-12-22; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Vancomycin
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vancomycin — adult patients treated with intravenous vancomycin in intensive care unit

SUMMARY:
The aim of this study was to assess factors that may influence vancomycin trough level and the rate achieving the target trough level in critically ill patients.

DETAILED DESCRIPTION:
This retrospective observational study included adult patients treated with intravenous vancomycin in intensive care unit of Zhongda Hospital from January 2015 to December 2017. Vancomycin dose was based on international consensus and adjusted according to estimated glomerular filtration rate (eGFR) calculated by the Cockcroft-Gault equation. vancomycin trough level (VTL) was retained at steady state (after the third dose). Linear regression was performed to determine the correlation between factors prior to the first vancomycin dose and VTL. Distribution of VTL and percentage of patients achieving the target trough level (15-20mg/L) was observed in different renal function.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients (age≥18 years) treated with intravenous vancomycin were included

Exclusion Criteria:

* Chronic renal dysfunction and acute renal injury patients treated with Renal Replacement therapy
* VTL was not retained at steady-state
* Vancomycin treatment time≤48h
* Vancomycin dose did not meet study definitions
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age≥18 years) treated with intravenous vancomycin were included. Exclusion criteria were chronic renal dysfunction and acute renal injury patients treated with Renal Replacement therapy, VTL was not retained at steady-state, vancomycin treatment time≤48h, vancomycin dose did not meet study definitions, palliative care.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients achieving the target vancomycin trough（15-20mg/L） | 3 years
  Vancomycin trough level was retained at steady state (after the third dose). If a patient has multiple measurements of vancomycin trough level, the first measurement is collected.Rate of patients achieving the target trough level (15-20mg/L) was observed.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, PHD., Principal Investigator — Southeast University